CLINICAL TRIAL: NCT01024127
Title: Genetic Predictors of AML Treatment Response
Brief Title: Studying DNA in Blood and Bone Marrow Samples From Younger Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B11; NCI-2011-02202 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000660540 (Other: Clinical Trials.gov); COG-AAML10B11 (Other: Children's Oncology Group); AAML10B11 (Other: Children's Oncology Group); AAML10B11 (Other: CTEP)
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood and bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-correlative (predictors of AML treatment outcomes): Germline DNA is obtained from previously collected peripheral blood or bone marrow samples for array-based genotyping studies, including genome-wide association studies (single nucleotide polymorphisms) and fine mapping genotyping. Clinical trial simulations are performed to test the clinical applicability of using genetic variation data in the management of infectious complications.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies deoxyribonucleic acid (DNA) in blood or bone marrow samples from younger patients with acute myeloid leukemia. Studying samples of blood and bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how well patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. Perform a genome-wide scan to test for loci associated with acute myeloid leukemia (AML) relapse and infection risk.

II. Validate positive associations seen in the genome-wide scan with a fine mapping approach.

III. Perform simulated clinical trials using germline genetic variation data to test the feasibility of using genetic data to inform the clinical care of pediatric patients with AML.

OUTLINE:

Germline DNA is obtained from previously collected peripheral blood or bone marrow samples for array-based genotyping studies, including genome-wide association studies (single nucleotide polymorphisms) and fine mapping genotyping. Clinical trial simulations are performed to test the clinical applicability of using genetic variation data in the management of infectious complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML

  * In remission
* Adequate DNA from peripheral blood or bone marrow samples
* Concurrent enrollment on CCG-2961, COG-AAML03P1, COG-AAML0531, AML-93, AML-97, AML-04,AML-09, or Canada AML Infection clinical trial required

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of AML in remission
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2009-12; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of first acute myeloid leukemia relapse | Up to 2 years
Rate of invasive bacterial infections defined as the number of invasive infection episodes divided by the days at risk | From study entry date to completion of therapy date provided on the final Reporting Period case reporting form, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aplenc, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Philadelphia, Pennsylvania, United States